CLINICAL TRIAL: NCT01033552
Title: MT2009-09: Biochemical Correction of Severe Epidermolysis Bullosa by Allogeneic Stem Cell Transplantation and "Off-the-shelf" Mesenchymal Stem Cells
Brief Title: Biochemical Correction of Severe EB by Allo HSCT and "Off-the-shelf" MSCs
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT2009-09; 0911M74035 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Antilymphocyte Serum; Mesenchymal Stem Cell Transplantation; Whole-Body Irradiation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- RDEB Mac (Experimental): Recessive Dystrophic EB (RDEB) - Myeloablative conditioning (MAC) Participants receive Myeloablative Busulfan (targeting AUC 1000 umol/min), Fludarabine 75 mg/m2, and Cyclophosphamide 200 mg/kg
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Myeloablative Busulfan; Procedure: Mesenchymal stem cell transplantation; Procedure: Bone marrow or umbilical cord blood (UCG) stem cell transplantation
- RDEB RIC (Experimental): Recessive Dystrophic EB (RDEB) - Reduced Intensity Condition Participants received Fludarabine 500 mg/m2, Cyclosphosphamide 50 mg/kg, equine Anti-thymocyte globulin 90 mg/kg, and low dose total body irradiation (either 200 or 300 cGy)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Anti-thymocyte globulin; Procedure: Mesenchymal stem cell transplantation; Radiation: Total body irradiation; Procedure: Bone marrow or umbilical cord blood (UCG) stem cell transplantation
- JEB MAC (Experimental): Junctional EB (JEB) - Myeloablative conditioning (MAC) Participants receive Myeloablative Busulfan (targeting AUC 1000 umol/min), Fludarabine 75 mg/m2, and Cyclophosphamide 200 mg/kg
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Myeloablative Busulfan; Procedure: Mesenchymal stem cell transplantation; Procedure: Bone marrow or umbilical cord blood (UCG) stem cell transplantation
- JEB RIC (Experimental): Junctional EB (JEB) - Reduced Intensity Condition Participants received Fludarabine 500 mg/m2, Cyclosphosphamide 50 mg/kg, equine Anti-thymocyte globulin 90 mg/kg, and low dose total body irradiation (either 200 or 300 cGy)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Anti-thymocyte globulin; Procedure: Mesenchymal stem cell transplantation; Radiation: Total body irradiation; Procedure: Bone marrow or umbilical cord blood (UCG) stem cell transplantation

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 50 mg/kg/day IV over 2 hours x 1 day, total dose 50 mg/kg will be administered on Day -6.
  Other Names: Cytoxan
Drug: Fludarabine — 40 mg/m^2/day intravenously on Days -6, -5, -4, -3 and -2.
  Other Names: Fludara
Drug: Anti-thymocyte globulin — 30 mg/kg on Days -4, -3 and -2.
  Other Names: ATG
  Arms: JEB RIC; RDEB RIC
Drug: Myeloablative Busulfan — Targeting AUC 1000 umol/min
  Arms: JEB MAC; RDEB Mac
Procedure: Mesenchymal stem cell transplantation — infused via intravenous drip on Day 0
  Other Names: MSCT
Radiation: Total body irradiation — 300 cGY on Day -1 administered in a single fraction at a dose rate of 10-19 cGy/minute prescribed to the midplane of the patient at the level of the umbilicus.
  Arms: JEB RIC; RDEB RIC
Procedure: Bone marrow or umbilical cord blood (UCG) stem cell transplantation — Bone marrow or UCB products will be infused as soon as the product arrives and within 30 minutes. The product is infused via IV drip.
  Other Names: UCBSCT

SUMMARY:
This is an open-label, single institution, phase II study in patients with epidermolysis bullosa (EB). The underlying hypothesis is that the infusion of bone marrow or umbilical cord blood from a healthy unaffected donor will correct the collagen, laminin, integrin, or plakin deficiency and reduce the skin fragility characteristic of severe forms of EB. A secondary hypothesis is that mesenchymal stem cells from a healthy donor will enhance the safety and efficacy of the allogeneic hematopoietic stem cell transplant as well as serve as a source of renewable cells for the treatment of focal areas of residual blistering.

DETAILED DESCRIPTION:
The primary objective of this study is to estimate the event-free survival rate by 1 year post-transplant with an event defined as a death or failure to have a demonstrable increase in collagen, laminin, integrin, keratin or plakin deposition by 1 year post-transplant or other biochemical, structural or physical measure of improvement.

The secondary objectives of this study are to i) determine the incidence of transplant-related mortality (TRM) at 180 days; ii) describe the pattern of biochemical improvement as measured by an increase in protein expression (collagen, laminin, integrin, keratin or plakin) and related structural and physical changes; iii) describe health quality of life at day 365 and 730 as compared to pretreatment results; iv) describe the pattern and durability of HSC and third party MSC engraftment in the skin; v) determine the probability of survival at 1 year.

Patients with severe epidermolysis bullosa will be screened to meet the eligibility requirements, related or unrelated donor marrow or UCB will be infused, and subjects will be followed for a minimum of 5 years after stem cell transplant. A target accrual of 75 subjects over 5 years will be recruited to the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe form of epidermolysis bullosa (EB) characterized by collagen, laminin, integrin, keratin or plakin deficiency. Assessment criteria for severe EB:

  * Documented collagen, laminin, integrin, keratin or plakin deficiency (by immunofluorescence staining with protein specific antibodies or Western blotting and by mutation analysis)
* Adequate Organ Function Criteria

  * Renal: glomerular filtration rate within normal range for age
  * Hepatic: bilirubin, aspartate aminotransferase/alanine aminotransferase (AST/ALT), Alkaline phosphatase (ALP) < 5 x upper limit of normal
  * Pulmonary: adequate pulmonary function in the opinion of the enrolling investigator
  * Cardiac: left ventricular ejection fraction ≥ 45%, normal electrocardiogram (EKG) or approved by Cardiology for transplant.
* Available Healthy HSC Donor (order of preference)

  * Related Donor (marrow or UCB)

    * HLA-A, B, C, DRB1 genotypic identical (sibling) donor
    * HLA-A, B, C, DRB1 phenotypic identical donor
    * 7/8 HLA matched donor at HLA-A, B, C, DRB1
  * Unrelated Donor

    * Marrow

      * HLA-A, B, C, DRB1 phenotypic identical donor
      * 7/8 HLA matched donor at HLA-A, B, C, DRB1
    * UCB

      * HLA-A, B (antigen level) and DRB1 (allele level) matched donor
      * 5/6 HLA matched donor at HLA-A, B, DRB1
      * 4/6 HLA matched donor at HLA-A, B, DRB1
* Voluntary written consent

Absence of Exclusion Criteria:

* Active systemic infection at time of transplantation (including active infection with Aspergillus or other mold within 30 days).
* History of human immunodeficiency virus (HIV) infection
* Evidence of squamous cell carcinoma
* Donor has EB
* Pregnancy females of child-bearing age must have a documented negative pregnancy test and agree to use contraception as a condition for enrollment.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Tolar, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center and Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC
Started | 7 | 16 | 2 | 7
Completed | 7 | 16 | 2 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC | Total
Number analyzed (Participants) | 7 | 16 | 2 | 7 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 15 | 2 | 7 | 31
  Between 18 and 65 years | 0 | 1 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 1 | 3 | 15
  Male | 4 | 8 | 1 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 6 | 15 | 2 | 5 | 28
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 7 | 9
  Asian | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 14 | 0 | 0 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 16 | 2 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Event-free Survival
Description: Event-free survival rate, with an event defined as death or failure to have a demonstrable increase in collagen, laminin, intergrin, keratin or plakin deposition. Assessed at follow up appointments through questionnaire and patient samples.
Time Frame: 1 year and 2 Years Post-transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC
Number analyzed (Participants) | 7 | 16 | 2 | 7
Percentage of participants
  1 year | 67 [19 to 90] | 80 [50 to 93] | 50 [1 to 91] | 29 [4 to 61]
  2 year | 44 [7 to 78] | 80 [50 to 93] | 50 [1 to 91] | 14 [1 to 46]

2. Secondary Outcome: Percentage of Participants Transplant-related Mortality (TRM)
Description: Incidence of transplant-related mortality (TRM)
Time Frame: 180 Days Post Transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC
Number analyzed (Participants) | 7 | 16 | 2 | 7
Percentage of participants | 43 [11 to 75] | 19 [2 to 36] | 50 [1 to 99] | 86 [50 to 100]

3. Secondary Outcome: Average Biochemical Improvement
Description: Pattern of biochemical improvement measured by cumulative increase in protein expression and related structural and physical changes
Time Frame: 1 Year Post-Transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC
Number analyzed (Participants) | 7 | 16 | 2 | 7
Percentage of participants | 29 [7 to 74] | 31 [14 to 60] | 0 [0 to 100] | 0 [0 to 100]

4. Secondary Outcome: Measure Patients Quality of Life Using a Questionnaire
Description: Health quality of life questionnaire as compared to pretreatment results. Scores can range from 0 to 100. The QOLS scores are summed so that a higher score indicates higher quality of life.
Time Frame: Pretreatment and 1 year
Population: Participants unnable to complete quality of life questionnaires at various time points.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC
Number analyzed (Participants) | 4 | 6 | 0 | 2
Scores on a scale
  Pretreatment | 43 [1 to 85] | 17 [1 to 79] |  | 1 [1 to 1]
  1 year: number analyzed (Participants) | 2 | 3 | 0 | 0
  1 year | 37 [1 to 79] | 68 [52 to 84] |  |

5. Secondary Outcome: Durability of HSC Donor Engraftment in the Skin
Description: Incidence of HSC donor engraftment in the skin
Time Frame: 100 Days
Measure: Number (95% Confidence Interval); unit: Percentage of Incidence
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC
Number analyzed (Participants) | 6 | 14 | 1 | 3
Percentage of Incidence | 11 [6 to 30] | 7 [0 to 18] | 0 [0 to 100] | 9 [0 to 13]

6. Secondary Outcome: Probability of Survival
Description: Surviving patients one year after engraftment
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC
Number analyzed (Participants) | 7 | 16 | 2 | 7
Percentage of participants | 71 [26 to 92] | 81 [52 to 94] | 50 [1 to 91] | 29 [4 to 61]

7. Secondary Outcome: Percentage of Participants Who Experienced Acute GVHD
Description: Incidence of acute GCHD
Time Frame: 100 Days
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC
Number analyzed (Participants) | 7 | 16 | 2 | 7
Percentage of participants | 14 [0 to 38] | 19 [0 to 37] | 0 [0 to 100] | 29 [0 to 60]

ADVERSE EVENTS:
Time Frame: 1 year through treatment
Arm/Group | RDEB Mac | RDEB RIC | JEB MAC | JEB RIC
All-Cause Mortality (participants affected / at risk) | 4/7 | 3/16 | 1/2 | 6/7
Serious Adverse Events (participants affected / at risk) | 7/7 | 16/16 | 2/2 | 7/7
Other Adverse Events (participants affected / at risk) | 7/7 | 16/16 | 2/2 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RDEB Mac (N=7) | RDEB RIC (N=16) | JEB MAC (N=2) | JEB RIC (N=7)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 3 (8) | 8 (11) | 0 (0) | 2 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 4 (4) | 6 (9) | 1 (2) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RDEB Mac (N=7) | RDEB RIC (N=16) | JEB MAC (N=2) | JEB RIC (N=7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (13) | 2 (2) | 0 (0) | 2 (3)
Chills (General disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 12 (25) | 2 (4) | 6 (12)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (6)
Rash (Skin and subcutaneous tissue disorders) | 7 (17) | 1 (1) | 2 (6) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 6 (14) | 10 (22) | 1 (2) | 6 (11)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders - Other (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT01033552/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT01033552/ICF_001.pdf